CLINICAL TRIAL: NCT00062504
Title: A Phase II Trial of Talampanel in Patients With Recurrent High-Grade Gliomas.
Brief Title: Phase 2 Trial Using Talampanel in Patients With Recurrent High Grade Gliomas
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Rivka Kreitman, Ph.D., Vice President, Innovative Research and Development, Teva Neuroscience
Model: Parallel | Purpose: Treatment
Other Study IDs: IXR-205-21-189
Record Dates: First submitted 2003-06-06; First posted 2003-06-12 (Estimated); Last update posted 2011-05-23 (Estimated); Status verified 2011-05

CONDITIONS: Glioblastoma Multiforme; Anaplastic Astrocytoma; Anaplastic Oligodendroglioma; Anaplastic Mixed Oligoastrocytoma
MeSH Terms: conditions — Glioblastoma; Astrocytoma; Oligodendroglioma | interventions — talampanel

ARMS (3):
- 1 (Experimental): Valproic: 10mg TID week 1, 25mg TID week 2, 35mg week 3
  Interventions: Drug: Talampanel
- 2 (Experimental): Non-enzyme-inducing anti-epileptic drugs: 25mg TID week 1, 35mg week 2, 50mg week 3
  Interventions: Drug: Talampanel
- 3 (Experimental): Enzyme-inducing anti-epileptic drugs: 35mg TID week 1, 505mg week 2, 75mg week 3
  Interventions: Drug: Talampanel

INTERVENTIONS:
Drug: Talampanel — 10mg, 25 mg, 35 mg, 50 mg, 75mg TID for 3 weeks

SUMMARY:
To analyze the effect of Talampanel on progression free survival in patients with recurrent high grade gliomas.

DETAILED DESCRIPTION:
To determine the efficacy of Talampanel in patients with recurrent malignant glioma as measured by 6-month progression survival, as well as to obtain preliminary information regarding the spectrum of toxicities of the drug among this patient population.

ELIGIBILITY:
Inclusion

1. Patients with histologically proven intracranial malignant glioma will be eligible for this protocol. Malignant glioma include glioblastoma multiforme (GBM), anaplastic astrocytoma (AA), anaplastic oligodendroglioma (AO), anaplastic mixed oligoastrocytoma (AMO), or malignant astrocytoma NOS (not otherwise specified).
2. Patients must have unequivocal evidence for tumor progression by MRI or CT scan. This scan should be performed within 14 days prior to registration and on a steroid dosage that has been stable for at least 5 days.
3. Patients having undergone recent resection of recurrent or progressive tumor will be eligible as long as all of the following conditions apply:

   1. They have recovered from the effects of surgery.
   2. Residual disease following resection of recurrent tumor is not mandated for eligibility into the study. To best assess the extent of residual disease post-operatively, a CT/ MRI should be done:

      * no later than 96 hours in the immediate post-operative period or
      * at least 4 weeks post-operatively, and
      * within 14 days of registration, and
      * on a steroid dosage that has been stable for at least 5 days.
4. If the 96-hour scan is more than 21 days before registration, the scan needs to be repeated.
5. Patients must have failed prior radiation therapy and must have an interval of greater than or equal to 4 weeks from the completion of radiation therapy to study entry.
6. All patients must sign an informed consent indicating that they are aware of the investigational nature of this study.
7. Patients must be > 18 years old, and with a life expectancy > 8 weeks.
8. Patients must have a Karnofsky performance status of > 60.
9. Patients must have recovered from the toxic effects of prior therapy: 4 weeks from any investigational agent, 4 weeks from prior cytotoxic therapy, two weeks from vincristine, 6 weeks from nitrosoureas, 3 weeks from procarbazine administration, and 1 week for non-cytotoxic agents, e.g., interferon, tamoxifen, thalidomide, cis-retinoic acid, etc. (radiosensitizer does not count).
10. Patients must have adequate bone marrow function (ANC > 1,200/mm3, platelet count of > 100,000/mm3, and hemoglobin > 10 gm/dl), adequate liver function (SGOT and bilirubin < 2 times ULN), and adequate renal function (serum creatinine < 1.5 mg/dL otherwise a measured 24-hour creatinine clearance > 60 cc/min) before starting therapy. These tests must be performed within 14 days prior to registration.
11. Patients must not have any significant medical illnesses that in the investigator's opinion cannot be adequately controlled with appropriate therapy or would compromise the patients' ability to tolerate this therapy.
12. This study was designed to include women and minorities, but was not designed to measure differences of intervention effects.
13. Patients must not have active infection requiring IV antibiotics.
14. Patients must not be pregnant or nursing, and all patients (both men and women) must be willing to practice birth control during and for 2 months after treatment with Talampanel. Women of childbearing potential (WCBP) must have a negative serum or urine pregnancy test. In addition, sexually active WCBP must agree to use adequate contraceptive methods (oral, injectable, or implantable hormonal contraceptive; tubal ligation; intra-uterine device; barrier contraceptive with spermicide; or vasectomized partner).

Exclusion Criteria

1. Patients who, in the view of the treating physician, have significant active cardiac, hepatic, renal, or psychiatric diseases are ineligible that would significantly increase the risk of using talampanel.
2. No concurrent use of other standard chemotherapeutics or investigative agents.
3. Patients known to have an active, life-threatening malignancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2003-07; Primary Completion 2006-01 (Actual); Study Completion 2006-04 (Actual)